CLINICAL TRIAL: NCT04592016
Title: A Single Center, Open-label, Clinical Study to Evaluate the Ability of Dermal Open Flow Microperfusion (dOFM) for Bioequivalence Testing of Topically Applied Diclofenac Sodium Products in Healthy Subjects
Brief Title: Evaluate the Ability of dOFM for BE Testing of Topically Applied Diclofenac Sodium Products in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joanneum Research Forschungsgesellschaft mbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: FDA02_Aim3; 2020-002101-25 (EudraCT Number)
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Dermal open flow microperfusion; Dermal Pharmacokinetics Measurement
MeSH Terms: interventions — halofantrine; Diclofenac; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilot Study (Experimental): Dermal-sampling visit: Measurement of dermal pharmacokinetic (PK) parameter (AUC, Cmax) of diclofenac using dermal open flow microperfusion (dOFM) after topical application of diclofenac sodium products in 6 participants. Additionally systemic appearance of diclofenac is measured by blood sampling.
  Interventions: Drug: Voltaren - Diclofenac sodium gel 1% (GSK, USA); Drug: Pennsaid 2 % Topical Solution (Horizon Therapeutics, USA); Device: Dermal open flow microperfusion - Pilot; Procedure: Blood sampling - Pilot
- Pivotal Study (Experimental): Dermal-sampling visit: Measurement of dermal pharmacokinetic (PK) parameter (AUC, Cmax) of diclofenac using dermal open flow microperfusion (dOFM) after topical application of diclofenac sodium products in 20 participants. Additionally systemic appearance of diclofenac is measured by blood sampling.
  Interventions: Drug: Voltaren - Diclofenac sodium gel 1% (GSK, USA); Drug: Pennsaid 2 % Topical Solution (Horizon Therapeutics, USA); Drug: Diclofenac sodium gel 1% (Perrigo, USA); Device: Dermal open flow microperfusion - Pivotal; Procedure: Blood sampling - Pivotal

INTERVENTIONS:
Drug: Voltaren - Diclofenac sodium gel 1% (GSK, USA) — Topical application in dermal-sampling visit
Drug: Pennsaid 2 % Topical Solution (Horizon Therapeutics, USA) — Topical application in dermal-sampling visit
Drug: Diclofenac sodium gel 1% (Perrigo, USA) — Topical application in dermal-sampling visit
  Arms: Pivotal Study
Device: Dermal open flow microperfusion - Pilot — Dermal open flow microperfusion will be used to collect interstitial fluid in order to assess diclofenac concentration in the dermis. Interstitial fluid (ISF) sampling: 1 hour pre-dose and 24 hours post-dose.
  Arms: Pilot Study
Device: Dermal open flow microperfusion - Pivotal — Dermal open flow microperfusion will be used to collect interstitial fluid in order to assess diclofenac concentration in the dermis. Interstitial fluid (ISF) sampling: 1 hour pre-dose and 12 hours post-dose.
  Arms: Pivotal Study
Procedure: Blood sampling - Pilot — 1 sample is taken pre-dose and 24 samples are taken post-dose.
  Arms: Pilot Study
Procedure: Blood sampling - Pivotal — 1 sample is taken pre-dose and 12 samples are taken post-dose.
  Arms: Pivotal Study

SUMMARY:
This will be a single center, open label, exploratory research study to assess the dermal pharmacokinetic (PK) profile of three marketed diclofenac products in 26 healthy volunteers using dermal open flow microperfusion (dOFM).

This clinical study aims to assess bioequivalence (BE) of three different diclofenac products.

DETAILED DESCRIPTION:
The clinical study is divided into a pilot and a pivotal study. The pilot study will involve 6 healthy adult volunteers. The pilot study aims to develop the optimal study design for the pivotal study by defining the dose of the reference product (diclofenac sodium gel 1%) and by evaluating the absence of significant systemic cross-talk (systemic redistribution) and lateral diffusion (cross-talk between adjacent treatment sites), which could increase background drug levels in the dermis that might confound the discrimination of dermal PK profiles between different products. Additionally, the suitability of a non-equivalent test product to serve as negative control for BE relative to the reference product will be evaluated.

The pivotal study will involve 20 healthy adult volunteers. In each volunteer the dermal PK profile of three different diclofenac products will be assessed in 6 topical treatment sites using dermal open flow microperfusion (dOFM), where the diclofenac penetration will be measured from baseline to 12 h post-dose. BE of the reference product against a generic test product (positive control) and against a non-equivalent test product (negative control) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult volunteers of age 18 to 65 years (both inclusive).
2. Males or non-pregnant, non-breast feeding females using adequate contraceptive methods or abstinence.
3. Able to read, understand and sign the written informed consent form.
4. Willing to follow the protocol requirements and comply with protocol restrictions.

Exclusion Criteria:

1. Social habits

   1. Smoker who is not willing to refrain from smoking during the in-house visit.
   2. History of drug and/or alcohol abuse within one year of start of study as judged by the investigator.
2. Medications: Use of any medications other than hormonal contraceptive, hormone replacement therapy or routine vitamins within the 7 days or 5 half-life periods whichever is longer prior to the initial dose of study medication.
3. Diseases: Presence of any clinically relevant acute or chronic disease, which in the investigator´s opinion might jeopardise subject's safety, evaluation of results or compliance with the protocol.
4. Any reason, which in the opinion of the investigator, would prevent the subject from safely participating in the study.
5. Any abnormalities found during physical examination or vital signs, unless deemed not clinically significant by the investigator.
6. Clinically significant abnormal laboratory evaluation results, as deemed by the investigator.
7. Clinically significant abnormal 12-lead ECG at screening, as deemed by the investigator.
8. Positive results to the test for hepatitis B antigen or hepatitis C antibodies.
9. Positive HIV test.
10. Positive alcohol breath test.
11. Blood donation within 30 days or significant loss of blood or plasma (more than 550 ml) within 90 days prior to screening.
12. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
13. Known hypersensitivity to diclofenac or any components of the drugs.
14. Tattoos or broken and/or damaged skin and/or scarring at the application areas.
15. Active skin diseases like psoriasis or atopic dermatitis, as judged by the investigator.
16. Subjects prone to keloid or hypertrophic scar formation or any known wound healing disorder.
17. Recent and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc.), as judged by the investigator.
18. Not willing to avoid excessive sun exposure, steam baths, sauna, swimming and other strenuous activities for 14 days after Visit 2 to ensure good tissue regeneration.
19. Not willing to refrain from shaving the planned treatment sites or using skin care products on the planned treatment sites for at least 5 days prior to start of Visit 2.
20. Pronounced hairiness on the planned treatment sites that may negatively affect BE testing.
21. Known allergy/hypersensitivity to any of the materials/supplies used during the study.
22. Presence of needle phobia.
23. Increased risk of thrombosis, e.g. personal or first degree relative(s) history of deep vein thrombosis.
24. Not enough space on the thighs for the dOFM probe set-up (minimum length of 24 cm, 3 treatment sites with 4 dOFM probes).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Area under the dermal concentration versus time curve for diclofenac (pilot study: 6 participants, pivotal study: 20 participants) | 25 hours (pilot study), 13 hours (pivotal study)
  Dermal concentrations (ng/mL) of diclofenac will be measured to calculate the area under the dermal concentration versus time curve AUC (ng*h/mL).
Maximal dermal concentration of diclofenac (pilot study: 6 participants, pivotal study: 20 participants) | 25 hours (pilot study), 13 hours (pivotal study)
  Dermal concentrations (ng/mL) of diclofenac will be measured to calculate the maximal dermal concentration (ng/mL).

SECONDARY OUTCOMES:
Blood diclofenac concentrations versus time curve (pilot study: 6 participants, pivotal study: 20 participants) | 25 hours (pilot study), 13 hours (pivotal study)
  Diclofenac concentrations (ng/mL) in the blood will be measured to obtain the concentration-time curves in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pieber, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- CTU - Clinical Trials Unit, Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bodenlenz M, Tiffner KI, Raml R, Augustin T, Dragatin C, Birngruber T, Schimek D, Schwagerle G, Pieber TR, Raney SG, Kanfer I, Sinner F. Open Flow Microperfusion as a Dermal Pharmacokinetic Approach to Evaluate Topical Bioequivalence. Clin Pharmacokinet. 2017 Jan;56(1):91-98. doi: 10.1007/s40262-016-0442-z. PMID 27539717
- [Background] Benfeldt E, Hansen SH, Volund A, Menne T, Shah VP. Bioequivalence of topical formulations in humans: evaluation by dermal microdialysis sampling and the dermatopharmacokinetic method. J Invest Dermatol. 2007 Jan;127(1):170-8. doi: 10.1038/sj.jid.5700495. Epub 2006 Jul 27. PMID 16874309
- [Background] Bodenlenz M, Aigner B, Dragatin C, Liebenberger L, Zahiragic S, Hofferer C, Birngruber T, Priedl J, Feichtner F, Schaupp L, Korsatko S, Ratzer M, Magnes C, Pieber TR, Sinner F. Clinical applicability of dOFM devices for dermal sampling. Skin Res Technol. 2013 Nov;19(4):474-83. doi: 10.1111/srt.12071. Epub 2013 Apr 13. PMID 23581539
- [Background] Bodenlenz M, Augustin T, Birngruber T, Tiffner KI, Boulgaropoulos B, Schwingenschuh S, Raney SG, Rantou E, Sinner F. Variability of Skin Pharmacokinetic Data: Insights from a Topical Bioequivalence Study Using Dermal Open Flow Microperfusion. Pharm Res. 2020 Sep 28;37(10):204. doi: 10.1007/s11095-020-02920-x. PMID 32989514
- [Background] Dehghanyar P, Mayer BX, Namiranian K, Mascher H, Muller M, Brunner M. Topical skin penetration of diclofenac after single- and multiple-dose application. Int J Clin Pharmacol Ther. 2004 Jul;42(7):353-9. doi: 10.5414/cpp42353. PMID 15605686
- [Background] Muller M, Mascher H, Kikuta C, Schafer S, Brunner M, Dorner G, Eichler HG. Diclofenac concentrations in defined tissue layers after topical administration. Clin Pharmacol Ther. 1997 Sep;62(3):293-9. doi: 10.1016/S0009-9236(97)90032-1. PMID 9333105